CLINICAL TRIAL: NCT04539483
Title: A Randomised, Double-Blind Phase II Trial of Topical HDIT101 Versus Placebo in Patients With Chronic Recurrent HSV-1 Infection and Orolabial Lesion
Brief Title: Monoclonal Antibody Therapy Against Chronic Herpes Simplex Virus 1 Infection
Acronym: MATCH-1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: stopped for futility in interim analysis
Sponsor: Heidelberg ImmunoTherapeutics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HTX101-03L
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Herpes Labialis
Keywords: Herpes simplex virus 1
MeSH Terms: conditions — Herpes Labialis | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HDIT101 (Experimental): Topical application of HDIT101 solution to orolabial herpes lesion (4 times over 2 days). Blinded study drug will be applied to 2 lesions in the study
  Interventions: Drug: HDIT101 (blinded therapy); Behavioral: Photo documentation of orolabial herpes lesions; Behavioral: Completion of questionnaires (patient-reported outcomes); Procedure: 28-day swabbing of orolabial region; Procedure: Blood drawings
- Placebo to HDIT101 (Placebo Comparator): Topical application of placebo solution to orolabial herpes lesion (4 times over 2 days). Blinded study drug will be applied to 2 lesions in the study
  Interventions: Drug: Placebo (blinded therapy); Behavioral: Photo documentation of orolabial herpes lesions; Behavioral: Completion of questionnaires (patient-reported outcomes); Procedure: 28-day swabbing of orolabial region; Procedure: Blood drawings

INTERVENTIONS:
Drug: HDIT101 (blinded therapy) — Patients will be treated with with topical HDIT101 (twice daily for 2 days). Blinded study drug will be applied to the first 2 lesions occuring in the treatment phase.
  Arms: HDIT101
Drug: Placebo (blinded therapy) — Patients will be treated with with topical placebo (twice daily for 2 days). Blinded study drug will be applied to the first 2 lesions occuring in the treatment phase.
  Arms: Placebo to HDIT101
Behavioral: Photo documentation of orolabial herpes lesions — Patients will be asked to document their orolabial lesions with photos by using their smart phone
Behavioral: Completion of questionnaires (patient-reported outcomes) — Patients will be asked to document their health status in questionnaires by using their smart phone
Procedure: 28-day swabbing of orolabial region — Patients will be asked to complete 3 episodes of 28-day swabbing of orolabial lesions
Procedure: Blood drawings — Blood will be drawn for e.g. safety lab, HSV-analysis, pharmacokinetic etc.

SUMMARY:
This is a phase II, double-blind, randomised, controlled, multicentre trial of topical HDIT101 versus placebo. HSV-1-positive patients with at least 6 orolabial herpes lesions in the last 12 months can be included.

The patients need to present with 3 herpes lesions within a 9 months observation phase. With the occurrence of the third lesion, the patients will enter the 12 months treatment phase and will be randomized in a 2:1 ratio to topical HDIT or placebo applied over 2 days. A potential fourth lesion will also be treated with the blinded study medication and additional lesions will be documented.

In a 12 months post-trial follow-up phase, further information on the occurence of lesions will be collected 4 times by phone.

Study duration per patient will be up to 21 months plus 12 months post-trial follow-up by phone. Patients need to come for study visits up to 9 times.

DETAILED DESCRIPTION:
This is a phase II, double-blind, randomised, controlled, multicentre trial of topical HDIT101 versus placebo.

Approximately 138 eligible patients will be randomised at a ratio of 2:1 to topical HDIT or corresponding placebo.

The trial consists of 3 parts: An observation phase (up to 9 months), a treatment phase of 12 months, and a post-trial follow-up phase of additional 12 months: The observation phase ensures that the patient develops a minimum number of lesions during the trial. In the 12 months treatment phase, blinded study treatment consisting of topical HDIT101 or placebo is applied to the patients at the first and second lesion episode. After completion of the treatment phase, patients are followed for additional 12 months for assessment of the development of further lesions (post-trial follow-up phase).

Observation phase (max. 9 months):

Eligible patients suffering from chronic recurrent herpes orolabialis for at least 12 months and reporting ≥ 6 lesions in the last 12 months can enter the observation phase. This part of the study serves for confirmation that patients develop a minimum number of 3 lesions within the 9 months observation period. No study treatment is applied in the observation phase, but standard-of-care treatment (SoC) can optionally be applied. Single swabs should additionally be taken from the lesion for confirmation of HSV-1 positivity.

Patients not developing 3 lesions with an HSV lesion score 3-7 during the 9 months observation phase are considered screening failures and will not be randomised into the treatment part of the trial.

Randomised, double-blind treatment phase (12 months):

This phase consists of four scheduled visits (day 30/120/240/365) and unscheduled visits for treatment of lesion 3 and 4, respectively.

Patients who have developed 3 outbreaks within the observational phase will enter the treatment phase. The third of these lesions will already be treated. Notably, patients do not have to complete the 9 months observation phase if they develop the 3rd lesion earlier - treatment starts with occurrence of a 3rd lesion.

With the occurrence of lesion 3 within the 9 months observation phase, patients need to schedule a visit at the study site when a vesicle is present. If the patient meets all inclusion criteria, randomisation takes place. An electronic patient reported outcome (ePRO) tool will be installed on the patients' devices and questionnaires will be answered. The lesion will be documented in the ePRO app with a photo. A swab of the lesion will be taken which preferably should contain fluid from the vesicular lesion. Subsequently, blinded IMP will be applied to the lesion. The investigator will determine the lesion start and end date based on information provided by the patient. 3 additional vials of study IMP for further treatment of this lesion will be handed over to the patient for self-application.

Upon occurrence of a fourth lesion in the treatment phase, the same procedure will be repeated at another unscheduled visit at the site when a vesicle is present. Again, IMP will be handed over to the patient for further treatment of this lesion.

All subsequent lesions occurring during the 12 months treatment phase need to be documented by the patient by photos and questionnaires. At each lesion episode, single swabs will be taken, but no further IMP will be applied and no unscheduled visit is necessary, but phone calls. The investigator will assess and medically confirm the lesion to be herpes-related and will determine the lesion start and end date based on information and photos provided by the patient and patient entries in the ePRO. Standard-of-care treatment (SoC) can optionally be applied.

Treatments and Examinations during the Study:

During all phases of the trial, patients need to report disease-specific symptoms and outbreak impact upon recognition of first symptoms during the study.

Orolabial viral shedding of patients is assessed by quantitative real time polymerase chain reaction (qRT-PCR) derived from swabs. These will be taken daily for 28 days in the orolabial region during the 9 months observation period starting after lesion 2, at occurrence of lesion 3 at visit 3 and 4 months after randomisation (starting at visit 5), respectively.

Each lesion recurrence has to be documented by the patient in the patient eDiary. In case of development of new lesions after lesion 3 or 4, patients will be instructed to take a swab of the lesion and provide this to the site for HSV-1 PCR outbreak confirmation. The patients must take photos (preferably daily) of the lesion until healing. These photos will be transferred to the sites' source data. The investigator will assess and medically confirm the lesion to be herpes-related and will determine the lesion start and end date based on information and photos provided by the patient and patient entries in the electronic diary.

Lesions will be rated according to a lesion score. For every lesion episode (outbreak), patients will be asked to report disease specific symptoms and outbreak impact in electronic questionnaires on a daily basis, from recognition of first symptoms until complete resolution of the symptoms.

Post-trial follow-up phase (12 months):

After the treatment phase, patients are further followed-up by phone every 3 months for a total duration of additional 12 months.

ELIGIBILITY:
Main Inclusion Criteria:

* Ability to provide written, personally signed and dated informed consent
* Age ≥ 18 years
* Understanding, ability, and willingness to fully comply with study interventions and restrictions.
* Seropositive for HSV-1 at screening with a history of chronic recurrent orolabial herpes infection for at least 12 months with at least 6 orolabial recurrences in the last year.
* Three confirmed lesions within 9 months after enrolment.
* Willingness not to use any HSV-suppressant therapy except 5% aciclovir cream as optional standard of care
* Willingness to remove beard or lip piercings if lesion boundaries in this region cannot be evaluated and topical treatment of the entire lesion is compromised (according to judgement of investigator).
* Willingness to self-obtain daily swabs from the orolabial region, to provide photos of the lesions and to complete questionnaires during the study.
* Medical assessment with no clinically significant morbidities or abnormalities as per judgement of the investigator.
* Willingness to use contraceptive methods for 30 days after each treatment.
* Availability of a mobile phone, tablet, or other smart device with a camera, connection to the internet and willingness to use this device for documentation of patient-reported outcomes and photo upload.

Main Exclusion Criteria:

* Patients who do not develop at least 3 lesions of stage 3 or higher during the 9 months observation phase or do not develop any lesion within 150 days from enrolment visit.
* Herpes keratitis.
* Requirement for immunosuppressive therapy and/or steroids.
* Any known clinically relevant allergies to drugs or any history of severe allergic or anaphylactic reactions
* Positive HIV antibody screen, active hepatitis B virus or active hepatitis C virus infection.
* Treatment with an investigational drug in any clinical study within the last 30 days prior to enrolment in this study.
* Prior treatment with HDIT101, e.g. in this or another clinical study.
* Prior vaccination with an HSV type 1/2 vaccine (e.g. experimental) within the last 2 years prior screening.
* Pregnant or breast-feeding women.
* Prior malignant disease (except basal cell carcinoma in situ) if not successfully cured more than 5 years before enrolment.
* Patients who have abnormal skin conditions which are considered clinically significant according to the assessment of the investigator
* Any clinically relevant medical history or current physical or psychiatric illnesses/medical conditions that constitute an unacceptable risk for study participation or make the participant unlikely to fully complete the study in the judgment of the investigator. This especially applies to currently medicated psychiatric illnesses since this poses an additional risk for pharmacodynamic interaction with IMP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 761 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Primary endpoint: Number of recurrences after topical HDIT101 versus placebo after 12 months. | During 12 months treatment phase
  The recurrence rate is defined as number of recurrences in the 12 months treatment phase divided by the total number of study days (in the 12 months treatment phase) after first IMP treatment

SECONDARY OUTCOMES:
Percentage of days with a lesion | During 12 months treatment phase
  Percentage of days with a lesion
Duration of recurrent lesions | During 12 months treatment phase
  Duration of recurrent lesions
Time to first recurrence | During 12 months treatment phase
  Time to first recurrence reported by the patient and verified by the investigator (If no further lesion develops, time to end of study is taken).
Number of aborted lesions | During 12 months treatment phase
  An aborted lesion is a non-ulcerative lesion that does not progress beyond the papule stage

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (5):
  - emovis GmbH, Berlin
  - Infektio Research GmbH & Co. KG, Frankfurt am Main
  - bioskin Prüfzentrum, Hamburg
  - ICH Study Center GmbH & Co. KG, Hamburg
  - Universitätsklinikum Heidelberg - Medizinische Klinik, Klinische Pharmakologie & Pharmakoepidemiologie, Heidelberg

IPD SHARING:
Plan to Share IPD: No